CLINICAL TRIAL: NCT00329017
Title: Correlation of SNP Patterns With Fine Needle Aspiration Cytomorphology in High Risk Postmenopausal Women
Brief Title: Protocol for Postmenopausal Women at Increased Risk of Developing Breast Cancer
Status: Withdrawn | Type: Observational
Why Stopped: No patients enrolled
Sponsor: Carol Fabian, MD (Other)
Collaborators: Intergenetics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Carol Fabian, MD, Professor, Director Breast Cancer Prevention Unit, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Other Study IDs: 9814
Record Dates: First submitted 2006-05-19; First posted 2006-05-24 (Estimated); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer
Keywords: SNPs; single nucleotide polymorphism; breast atypia; breast epithelial hyperplasia; high risk for breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fine needle aspirate
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Post-menopausal women who are at increased risk for development of breast cancer on the basis of family or personal history.
  Interventions: Procedure: Fine needle aspiration

INTERVENTIONS:
Procedure: Fine needle aspiration — Fine needle aspiration

SUMMARY:
A study to examine the potential associations between common single nucleotide polymorphisms and pre-cancerous conditions in breast tissue specimens from postmenopausal women.

DETAILED DESCRIPTION:
A study to examine the correlation between single nucleotide polymorphisms (SNPs) affecting steroid and carcinogen metabolism and benign breast tissue cytomorphology collected via random periareolar fine needle aspiration in postmenopausal women at increased risk for breast cancer and taking hormone replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women on or off hormone replacement therapy
* at high risk of developing breast cancer determined by family or personal history
* postmenopausal women not on hormone replacement therapy for at minimum six months prior to corresponding aspiration
* willing to participate in companion protocol (KUMC HSC#4601) for random periareolar fine needle aspiration (RPFNA) for correlational studies

Exclusion Criteria:

* women who have been on raloxifene, tamoxifen, letrozole, anastrozole or exemestane within the six months prior to RPFNA.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post menopausal women, on or off hormone replacement therapy, at high risk of developing breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-05; Primary Completion 2015-11-12 (Actual); Study Completion 2015-11-12 (Actual)

PRIMARY OUTCOMES:
Correlation of SNP patterns with cytlomorphology of breast fine needle aspirates. | ongoing
  develoment of algorithm for prediction of risk of developing breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Carol J Fabian, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
Global results will be published.